CLINICAL TRIAL: NCT07183514
Title: Clinical and Radiographic Evaluation of Eggshell-derived Calcium Hydroxyapatite Verses Calcium Hydroxide as In-direct Pulp Capping Agent in Permanent Molars
Brief Title: A Study Comparing Eggshell Based and Gold Standard Materials to Heal Deep Tooth Damage in Adult Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Arooj fatima, Post- graduate trainee in operative dentistry department PGMI Lahore, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGMI-LHR-2024-59
Record Dates: First submitted 2025-09-08; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Indirect Pulp Cap
Keywords: dental caries, indirect pulp capping, hydroxyapatite, reparative dentine
MeSH Terms: conditions — Dental Caries; Dentin, Secondary | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eggshell-derived calcium hydroxyapatite (Experimental): Participants in this arm will receive indirect pulp capping with eggshell-derived calcium hydroxyapatite, followed by restoration with glass ionomer cement and composite resin.
  Interventions: Biological: eggshell-derived calcium hydroxyapatite
- Calcium hydroxide (Active Comparator): Participants in this arm will receive indirect pulp capping with Calcium hydroxide, followed by restoration with glass ionomer cement and composite resin.
  Interventions: Biological: Calcium hydroxide

INTERVENTIONS:
Biological: eggshell-derived calcium hydroxyapatite — eggshell-derived calcium hydroxyapatite will be placed as an indirect pulp capping material after chemo-mechanical caries removal and before final restoration with glass ionomer cement and composite resin.
  Arms: eggshell-derived calcium hydroxyapatite
Biological: Calcium hydroxide — Calcium hydroxide will be placed as an indirect pulp capping material after chemo-mechanical caries removal and before final restoration with glass ionomer cement and composite resin.
  Arms: Calcium hydroxide

SUMMARY:
This clinical trial will evaluate the effectiveness of eggshell-derived calcium hydroxyapatite compared to calcium hydroxide as indirect pulp capping agent in permanent teeth. A total of 54 teeth from healthy individuals aged 18 to 40 years will be randomly allocated into two groups:

Group A (experimental) treated with eggshell-derived calcium hydroxyapatite. Group B (control) treated with calcium hydroxide.

After caries removal the assigned pulp capping agent will be applied, and the teeth will be restored. Clinical and radiographic evaluations will be performed at 1 and 3 months to assess pulp vitality, symptom-free status, and periapical health.

DETAILED DESCRIPTION:
Dental caries is the most prevalent bacterial disease affecting both primary and permanent dentition. Modern dental practice emphasizes minimally invasive techniques that preserve pulp vitality. Indirect pulp capping is one such procedure, performed in teeth without signs of irreversible pulpitis, where infected dentine is removed while caries-affected dentine (CAD) is preserved and covered with a biocompatible material.

Calcium hydroxide remains the most widely used pulp capping material despite its shortcomings. Hydroxyapatite, a stable synthetic calcium phosphate ceramic, has demonstrated excellent biocompatibility. Eggshells are a natural, abundant source of calcium carbonates and oxides, making them a promising precursor for hydroxyapatite.

This randomized, double-blind clinical trial aims to evaluate and compare the clinical and radiographic outcomes of eggshell-derived calcium hydroxyapatite and calcium hydroxide as indirect pulp capping agents in permanent teeth with deep caries. Fifty-four teeth from healthy individuals aged 18-40 will be included. Random allocation will be performed using the lottery method.

Group A (experimental) will receive eggshell-derived calcium hydroxyapatite, while Group B (control) will receive calcium hydroxide. Following rubber dam isolation and chemo-mechanical caries removal with carie-fix gel, infected dentine will be removed using a spoon excavator while CAD is preserved. The allocated pulp capping agent will be placed over CAD, followed by restoration with glass ionomer cement (GC Gold Label II) and composite resin.

Clinical and radiographic assessments will be carried out at 1 month and 3 months. Clinical evaluation will include pulp vitality, pain on percussion, and mobility. Radiographic assessment will include reparative dentine thickness and absence of periapical pathology.

The findings will determine whether eggshell-derived calcium hydroxyapatite can be considered a viable natural alternative to calcium hydroxide for indirect pulp capping.

ELIGIBILITY:
Inclusion Criteria:

1. Teeth with symptoms of reversible pulpitis.
2. Teeth that show positive response on electric pulp testing (EPT).
3. Teeth with caries penetrating up to three-quarters (¾) of dentine without pulp involvement.
4. Healthy cooperative patients of both sexes between 18 to 40 years of age.

   -

Exclusion Criteria:

1. Necrosed Teeth with radiolucency in the periapical and furcation regions.
2. Tooth with internal and external root resorption.
3. Periodontally compromised tooth. (BPE score 3 and above)
4. Physically and mentally handicapped patients. (ASA score 3 and above)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
clinical symptoms (pain on percussion, tooth mobility) and radiographic evaluation | 3 months
  Evaluates absence of pain and pathological mobility, Measures dentine bridge thickness and absence of periapical pathology.

SECONDARY OUTCOMES:
restoration success, post operative sensitivity | baseline to seven days
  Records patient-reported sensitivity and discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- de'Montmorency college of dentistry Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swarup JS, Thomas R, Rucharitha J, Arunkumar VR, V V. Eggshell-derived hydroxyapatite as a biomaterial in dentistry: a scoping review of synthesis, properties and applications. Evid Based Dent. 2025 Sep;26(3):153. doi: 10.1038/s41432-025-01146-3. Epub 2025 May 12. PMID 40355679
- [Background] Reddy, S.P. et al. (2020a) 'Clinical comparison of eggshell derived calcium hydroxyapatite with Dycal® as indirect pulp capping agents in primary molars', Pesquisa Brasileira em Odontopediatria e Clínica Integrada, 20.(e0041):1-9 doi:10.1590/pboci.2020.151.
- See also: A randomized clinical study comparing eggshell-derived calcium hydroxyapatite with Dycal® (calcium hydroxide) for indirect pulp capping in primary molars. The eggshell-derived hydroxyapatite group showed significantly greater reparative dentine formation — http://dx.doi.org/10.1590/pboci.2020.151
- See also: A scoping review covering synthesis, properties, and dental applications of eggshell-derived hydroxyapatite (E-HAp), including its use in pulp capping and regenerative endodontics. Provides comprehensive background on E-HAp's potential in dentistry — https://doi.org/10.1038/s41432-025-01146-3